CLINICAL TRIAL: NCT07345884
Title: Comparison of Treatment of Severe Acute Malnutrition in Children 6 to 59 Months Old With Standard Ready To Use Therapeutic Food and Newly Formulated Lipid Optimized Ready To Use Therapeutic Food an Individual Randomized Double Blind Controlled Trial
Brief Title: Treatment of Severe Acute Malnutrition in Children 6 to 59 Months Old With Standard Ready To Use Therapeutic Food Compared to a Newly Formulated Lipid Optimized Ready To Use Therapeutic Food
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ahmed Moutwakil, Co-Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-25-1096
Record Dates: First submitted 2026-01-02; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Severe Acute Malnutrition in Childhood; Malnutrition, Child; Neurocognition, Child
Keywords: RUTF; Ready-to-use therapeutic food
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Participants in both interventions will receive approximately 190 kcal/kg/day of LO-RUTF or standard RUTF. The standard RUTF will be produced internationally and shipped to Pakistan. The alternative treatment for SAM, LO-RUTF, is produced locally in Pakistan.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LO-RUTF (Experimental): Participants in the LO-RUTF arm will receive approximately 190 kcal/kg/day of Lipid-Optimized Ready to Use Therapeutic Food (RUTF). This RUTF is locally produced and contains maize, milk powder, rice flour, soymeal, sugar, whey isolate, palm oil, flaxseed oil, coconut oil, premix and an emulsifier.
  Interventions: Dietary Supplement: Lipid-Optimized Ready to Use Therapeutic Food (RUTF)
- RUTF (Active Comparator): Participants in the RUTF arm will receive approximately 190 kcal/kg/day of Ready to Use Therapeutic Food (RUTF). This RUTF produced by UNICEF contains peanut paste, sugar, non-fat dried milk, vegetable oil, a premix containing concentrated minerals and vitamins, and an emulsifier.
  Interventions: Dietary Supplement: Ready to Use Therapeutic Food (RUTF)

INTERVENTIONS:
Dietary Supplement: Lipid-Optimized Ready to Use Therapeutic Food (RUTF) — Since this is a pilot trial for the study recipe, we have increased the vitamin D3 content in this RUTF as an experimental variable within this study.
  Arms: LO-RUTF
Dietary Supplement: Ready to Use Therapeutic Food (RUTF) — This is the standard of care RUTF with UNICEF product specifications. This RUTF will be produced internationally and shipped to Pakistan.
  Other Names: UNICEF RUTF; Standard RUTF
  Arms: RUTF

SUMMARY:
The goal of this randomized clinical trial is to learn if a newly formulated Lipid-Optimized Ready-to-Use Therapeutic Food (LO-RUTF) can treat severe acute malnutrition in children aged 6 to 59 months. The main questions it aims to answer are:

1. Does LO-RUTF impact physical recovery from severe acute malnutrition in participants?
2. Does LO-RUTF impact neurocognitive performance after 8 and 12 weeks of treatment?

Researchers will compare LO-RUTF to standard RUTF see if our energy-dense food compares to standard issue RUTF in terms of promoting recovery from severe acute malnutrition.

Participants will

* Take a one-week ration of LO-RUTF or standard RUTF based on the participant's weight
* Return every week for checkups, tests and to receive the next ration of assigned RUTF if eligible
* Be assessed for neurocognitive function through Malawi Developmental Assessment Tool (MDAT) at three time points (before treatment, 4 weeks, 8 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-59 months with severe acute malnutrition, i.e., MUAC <11.5 cm, and/or weight-for-height/length z-score < -3, and/or with bilateral pitting edema, with an appetite to completely consume a 30 g test feeding, and without medical complications presenting at selected rural therapeutic feeding health facilities

Exclusion Criteria:

* Children that are simultaneously involved in another research trial or supplemental feeding program, are developmentally delayed, have vision or hearing deficits, or have a history of milk or peanut allergy.
* Chronic diseases such as malabsorption, chronic kidney disease, inflammatory bowel disease, congenital heart disease, endocrine disorders (e.g., hypothyroidism, growth hormone deficiencies), recurrent infections (e.g., pneumonia, cough, fever, pharyngitis), chronic respiratory diseases (e.g., asthma, lung diseases), congenital or acquired immunodeficiency, and neurological disorders

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Recovered from Severe Acute Malnutrition as Assessed by WHO Anthro v3.1 | From enrollment to the end of treatment at 8 weeks
  The primary outcome is recovery from SAM, deﬁned as: mid-upper arm circumference ≥ 11.5cm (for two consecutive weekly visits), and/or weight-for-height/length z-score > -3 SD, and/or no bilateral pitting edema (for two consecutive weekly visits).

SECONDARY OUTCOMES:
Change in MDAT Scores after 8 and 12 weeks of treatment | Baseline and after 8 and 12 weeks of treatment
  The global development score along with all subdomain scores of the MDAT will be used as a measure of neurocognitive performance. with a higher score indicating a better outcome.
Time to Recovery from Severe Acute Malnutrition | From enrollment to the end of the study period at 12 weeks
  Defined as time taken to recover from severe acute malnutrition, which is deﬁned as: mid-upper-arm-circumference ≥ 11.5cm (for two consecutive weekly visits), and/or weight-for-height z-score > -3, and/or no bilateral pitting edema (for two consecutive weekly visits).
Time to Recovery from Moderate Acute Malnutrition | From enrollment to the end of the study period at 12 weeks
  Defined as time taken to achieve a mid-upper-arm-circumference ≥12.5 cm
Proportion of Participants with Relapse of Moderate Acute Malnutrition | From enrollment to the end of the study period at 12 weeks
  Participants developing moderate acute malnutrition at any point after achieving recovery from severe acute malnutrition compared to all participants
Proportion of Participants with Relapse of Severe Acute Malnutrition | From enrollment to the end of the study period at 12 weeks
  Participants developing severe acute malnutrition at any point after achieving recovery from severe acute malnutrition compared to all participants
Number of Participants with Non-Responder Status | From enrollment to the end of the study period at 12 weeks
  Participants who have not met the SAM exit criteria after 3 months (MUAC > 11.5 cm, clinically well, > 15 % weight gain, and no oedema for two consecutive visits) will receive a non-responder outcome.
Incidence of Adverse Events | From enrollment to the end of the study period at 12 weeks
  Number of participants with any adverse events, including those judged to be related to the study RUTF
Incidence of Hypercalcemia, Hypervitaminosis D, or excessive DHA concentrations | From baseline to the end of treatment at 8 weeks
  Determined by biochemical assessments at 8 weeks to evaluate serum 25-hydroxyvitamin D, calcium, and DHA concentrations.

OTHER OUTCOMES:
Mortality rate of participants | From enrollment to the end of study period at 12 weeks
  Frequency of deaths among participants within study period

CONTACTS AND LOCATIONS:
Overall Officials: Kiran K Masood, MD, Principal Investigator — University of California, Los Angeles; Mohid Khan, Study Director — The Satya Nutrition Foundation; Samir Ismail, Study Chair — The Satya Nutrition Foundation; Akhila Annadanam, Study Chair — The Satya Nutrition Foundation; Tu Nguyen, Study Chair — The Satya Nutrition Foundation; Fatima Ahmad, Study Chair — The Satya Nutrition Foundation; Meghana Dantuluri, Study Chair — The Satya Nutrition Foundation; Amith Umesh, Study Director — The Satya Nutrition Foundation
Locations (1):
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes